CLINICAL TRIAL: NCT01327625
Title: A Pilot Study Evaluating the Efficacy of Azithromycin, N-acetylcystein and Inhaled Corticosteroid Combination Therapy for Bronchiolitis Obliterans After Allogeneic Hematopoietic Cell Transpantation
Brief Title: Efficacy Study of Azithromycin-based Therapy for Bronchiolitis Obliterans
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Preliminary reports of this study was too bad.
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Dae-Young Kim, Assistant Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-ALLO-041
Record Dates: First submitted 2011-03-31; First posted 2011-04-01 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Graft vs Host Disease; Bronchiolitis Obliterans
Keywords: Allogeneic hematopoietic cell transplantation; Graft versus host disease; Bronchiolitis obliterans; Azithromycin; N-acetylcystein; Fluticasone; Inhaled steroid
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans | interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azithromycin (Experimental): Patient who are diagnosed as bronchiolitis obliterans according to the WHO criteria
  Interventions: Drug: azithromycin + N-acetylcystein + inhaled corticosteroid

INTERVENTIONS:
Drug: azithromycin + N-acetylcystein + inhaled corticosteroid — * Azithromycin 500mg qd x 1 week --> 250mg qod x 6 months
  * N-acetylcystein 200mg tid x 6 months
  * Fluticasone 250mcg puff x2/day x 6 months
  Other Names: Zithromax

SUMMARY:
[Study Objectives]

* To evaluate the efficacy of azithromycin, N-acetylcystein, and inhaled corticosteroid combination therapy in patients with bronchiolitis obliterans as a complication of allogeneic hematopoietic cell transplantation in terms of response rate at 6 months after treatment initiation based on the improvement of FEV1.

DETAILED DESCRIPTION:
* Bronchiolitis obliterans (BO) is a graft-versus-host disease of respiratory organs.
* Prognosis of BO is very poor, and the overall outcome of patients who are involved in BO is very dismal.
* The mechanism of BO has been known to be associated with immune / non-immune response.
* Corticosteroid and immunosuppressants are recommended as a best current treatment options for BO, which have been not satisfactory.
* Many treatment options have been tried to improve the outcome of BO.
* Azithromycin, as an immune modulating agent, has been tried for the treatment of BO, and has been reported to show hopeful results.
* N-acetylcystein, as an antioxidative agent, has been tried for BO.
* Inhaled corticosteroid may help to improve airway inflammation and decrease the amount of systemic corticosteroid.
* These 3 drugs are widely used for other respiratory disease, have been proven to be safe, and have shown some efficacy for BO in various depth of evidence.
* In these rationale, we'd like to try the 3-drug combination for BO, to assess the efficacy and safety of these drug combination.

ELIGIBILITY:
Inclusion Criteria:

* Patients who previously received allogeneic hematopoietic cell transplantation due to hematologic malignancy, bone marrow failure syndrome, and other compatible disease.
* Patients who are diagnosed as bronchiolitis obliterans (BO) according to the NIH diagnostic guideline which is suggested as below.
* Patients should be 15 years of age or older, but younger than 75 years.
* Patients should have estimated life expectancy of more than 3 months.
* Patients must have adequate hepatic function (bilirubin less than 3.0 ㎎/㎗, AST and ALT less than three times the upper normal limit).
* Patients must have adequate renal function (creatinine less than 2.0 ㎎/㎗).

Exclusion Criteria:

* Presence of significant active infection
* Presence of uncontrolled bleeding
* Any coexisting major illness or organ failure
* Patients with a psychiatric disorder or mental deficiency severe as to make compliance with the treatment unlike, and making informed consent impossible.
* Nursing women, pregnant women, women of childbearing potential who do not want adequate contraception
* Patients with a diagnosis of prior malignancy unless disease-free for at least 5 years following therapy with curative intent (except curatively treated nonmelanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia)

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Response rate based on the improvement of FEV1 | 6 months
  Response rate at 6 months after treatment initiation based on the improvement of FEV1

SECONDARY OUTCOMES:
Clinical benefit rate based on the degree of change in FEV1 | 6 months
  Clinical benefit rate at 6 months after treatment initiation based on the degree of change in FEV1
change in FEV1 compared with pretreatment level | 6 months after treatment initiation
  Change in FEV1 at 6 months after treatment initiation compared with pretreatment level
Reduction rate in immunosuppressive agent / systemic corticosteroid | 6 months after treatment initiation
  Reduction rate in immunosuppressive agent / systemic corticosteroid at 6 months after treatment initiation
Discontinuation rate in immunosuppressive agent / systemic corticosteroid | 6 months after treatment initiation
  Discontinuation rate in immunosuppressive agent / systemic corticosteroid at 6 months after treatment initiation
Change in dose-intensity of immunosuppressive agent / systemic corticosteroid compared with pretreatment dose-intensity | 6 months after treatment initiation
  Change in dose-intensity of immunosuppressive agent / systemic corticosteroid at 6 month after treatment initiation compared with pretreatment dose-intensity
event-free survival | 1 year
overall survival | 1year

CONTACTS AND LOCATIONS:
Overall Officials: Dae-Young Kim, M.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Patriarca F, Poletti V, Costabel U, Battista ML, Sperotto A, Medeot M, Toffoletti E, Fanin R. Clinical presentation, outcome and risk factors of late-onset non-infectious pulmonary complications after allogeneic stem cell transplantation. Curr Stem Cell Res Ther. 2009 May;4(2):161-7. doi: 10.2174/157488809788167436. PMID 19442201
- [Background] Afessa B, Peters SG. Major complications following hematopoietic stem cell transplantation. Semin Respir Crit Care Med. 2006 Jun;27(3):297-309. doi: 10.1055/s-2006-945530. PMID 16791762
- [Background] Nishio N, Yagasaki H, Takahashi Y, Muramatsu H, Hama A, Tanaka M, Yoshida N, Watanabe N, Kudo K, Yoshimi A, Kojima S. Late-onset non-infectious pulmonary complications following allogeneic hematopoietic stem cell transplantation in children. Bone Marrow Transplant. 2009 Sep;44(5):303-8. doi: 10.1038/bmt.2009.33. Epub 2009 Apr 6. PMID 19349954
- [Background] Williams KM, Chien JW, Gladwin MT, Pavletic SZ. Bronchiolitis obliterans after allogeneic hematopoietic stem cell transplantation. JAMA. 2009 Jul 15;302(3):306-14. doi: 10.1001/jama.2009.1018. PMID 19602690
- [Background] Sato M, Keshavjee S. Bronchiolitis obliterans syndrome: alloimmune-dependent and -independent injury with aberrant tissue remodeling. Semin Thorac Cardiovasc Surg. 2008 Summer;20(2):173-82. doi: 10.1053/j.semtcvs.2008.05.002. PMID 18707652
- [Background] Duncan CN, Buonanno MR, Barry EV, Myers K, Peritz D, Lehmann L. Bronchiolitis obliterans following pediatric allogeneic hematopoietic stem cell transplantation. Bone Marrow Transplant. 2008 Jun;41(11):971-5. doi: 10.1038/bmt.2008.19. Epub 2008 Feb 25. PMID 18297116
- [Background] Ditschkowski M, Elmaagacli AH, Trenschel R, Peceny R, Koldehoff M, Schulte C, Beelen DW. T-cell depletion prevents from bronchiolitis obliterans and bronchiolitis obliterans with organizing pneumonia after allogeneic hematopoietic stem cell transplantation with related donors. Haematologica. 2007 Apr;92(4):558-61. doi: 10.3324/haematol.10710. PMID 17488669
- [Background] Huisman C, van der Straaten HM, Canninga-van Dijk MR, Fijnheer R, Verdonck LF. Pulmonary complications after T-cell-depleted allogeneic stem cell transplantation: low incidence and strong association with acute graft-versus-host disease. Bone Marrow Transplant. 2006 Oct;38(8):561-6. doi: 10.1038/sj.bmt.1705484. Epub 2006 Sep 4. PMID 16953211
- [Background] Yoshihara S, Tateishi U, Ando T, Kunitoh H, Suyama H, Onishi Y, Tanosaki R, Mineishi S. Lower incidence of Bronchiolitis obliterans in allogeneic hematopoietic stem cell transplantation with reduced-intensity conditioning compared with myeloablative conditioning. Bone Marrow Transplant. 2005 Jun;35(12):1195-200. doi: 10.1038/sj.bmt.1704985. PMID 15852024
- [Background] Santo Tomas LH, Loberiza FR Jr, Klein JP, Layde PM, Lipchik RJ, Rizzo JD, Bredeson CN, Horowitz MM. Risk factors for bronchiolitis obliterans in allogeneic hematopoietic stem-cell transplantation for leukemia. Chest. 2005 Jul;128(1):153-61. doi: 10.1378/chest.128.1.153. PMID 16002929
- [Background] Xu J, Torres E, Mora AL, Shim H, Ramirez A, Neujahr D, Brigham KL, Rojas M. Attenuation of obliterative bronchiolitis by a CXCR4 antagonist in the murine heterotopic tracheal transplant model. J Heart Lung Transplant. 2008 Dec;27(12):1302-10. doi: 10.1016/j.healun.2008.08.010. PMID 19059110
- [Background] Hildebrandt GC, Granell M, Urbano-Ispizua A, Wolff D, Hertenstein B, Greinix HT, Brenmoehl J, Schulz C, Dickinson AM, Hahn J, Rogler G, Andreesen R, Holler E. Recipient NOD2/CARD15 variants: a novel independent risk factor for the development of bronchiolitis obliterans after allogeneic stem cell transplantation. Biol Blood Marrow Transplant. 2008 Jan;14(1):67-74. doi: 10.1016/j.bbmt.2007.09.009. PMID 18158963
- [Background] Medoff BD, Wain JC, Seung E, Jackobek R, Means TK, Ginns LC, Farber JM, Luster AD. CXCR3 and its ligands in a murine model of obliterative bronchiolitis: regulation and function. J Immunol. 2006 Jun 1;176(11):7087-95. doi: 10.4049/jimmunol.176.11.7087. PMID 16709871
- [Background] Jaramillo A, Smith CR, Maruyama T, Zhang L, Patterson GA, Mohanakumar T. Anti-HLA class I antibody binding to airway epithelial cells induces production of fibrogenic growth factors and apoptotic cell death: a possible mechanism for bronchiolitis obliterans syndrome. Hum Immunol. 2003 May;64(5):521-9. doi: 10.1016/s0198-8859(03)00038-7. PMID 12691702
- [Background] Belperio JA, DiGiovine B, Keane MP, Burdick MD, Ying Xue Y, Ross DJ, Lynch JP 3rd, Kunkel SL, Strieter RM. Interleukin-1 receptor antagonist as a biomarker for bronchiolitis obliterans syndrome in lung transplant recipients. Transplantation. 2002 Feb 27;73(4):591-9. doi: 10.1097/00007890-200202270-00020. PMID 11889437
- [Background] Belperio JA, Keane MP, Burdick MD, Lynch JP 3rd, Xue YY, Berlin A, Ross DJ, Kunkel SL, Charo IF, Strieter RM. Critical role for the chemokine MCP-1/CCR2 in the pathogenesis of bronchiolitis obliterans syndrome. J Clin Invest. 2001 Aug;108(4):547-56. doi: 10.1172/JCI12214. PMID 11518728
- [Background] Vilchez RA, Dauber J, Kusne S. Infectious etiology of bronchiolitis obliterans: the respiratory viruses connection - myth or reality? Am J Transplant. 2003 Mar;3(3):245-9. doi: 10.1034/j.1600-6143.2003.00056.x. PMID 12614277
- [Background] Dudek AZ, Mahaseth H, DeFor TE, Weisdorf DJ. Bronchiolitis obliterans in chronic graft-versus-host disease: analysis of risk factors and treatment outcomes. Biol Blood Marrow Transplant. 2003 Oct;9(10):657-66. doi: 10.1016/s1083-8791(03)00242-8. PMID 14569562
- [Background] Chien JW, Duncan S, Williams KM, Pavletic SZ. Bronchiolitis obliterans syndrome after allogeneic hematopoietic stem cell transplantation-an increasingly recognized manifestation of chronic graft-versus-host disease. Biol Blood Marrow Transplant. 2010 Jan;16(1 Suppl):S106-14. doi: 10.1016/j.bbmt.2009.11.002. Epub 2009 Nov 5. PMID 19896545
- [Background] Maimon N, Lipton JH, Chan CK, Marras TK. Macrolides in the treatment of bronchiolitis obliterans in allograft recipients. Bone Marrow Transplant. 2009 Jul;44(2):69-73. doi: 10.1038/bmt.2009.106. Epub 2009 May 11. PMID 19430505
- [Background] Gottlieb J, Szangolies J, Koehnlein T, Golpon H, Simon A, Welte T. Long-term azithromycin for bronchiolitis obliterans syndrome after lung transplantation. Transplantation. 2008 Jan 15;85(1):36-41. doi: 10.1097/01.tp.0000295981.84633.bc. PMID 18192909
- [Background] Verleden GM, Dupont LJ. Azithromycin therapy for patients with bronchiolitis obliterans syndrome after lung transplantation. Transplantation. 2004 May 15;77(9):1465-7. doi: 10.1097/01.tp.0000122412.80864.43. PMID 15167610
- [Background] Khalid M, Al Saghir A, Saleemi S, Al Dammas S, Zeitouni M, Al Mobeireek A, Chaudhry N, Sahovic E. Azithromycin in bronchiolitis obliterans complicating bone marrow transplantation: a preliminary study. Eur Respir J. 2005 Mar;25(3):490-3. doi: 10.1183/09031936.05.00020804. PMID 15738293
- [Background] Meloni F, Cascina A, Miserere S, Perotti C, Vitulo P, Fietta AM. Peripheral CD4(+)CD25(+) TREG cell counts and the response to extracorporeal photopheresis in lung transplant recipients. Transplant Proc. 2007 Jan-Feb;39(1):213-7. doi: 10.1016/j.transproceed.2006.10.227. PMID 17275508
- [Background] Duncan CN, Barry EV, Lehmann LE. Tolerability of pravastatin in pediatric hematopoietic stem cell transplant patients with bronchiolitis obliterans. J Pediatr Hematol Oncol. 2010 Apr;32(3):185-8. doi: 10.1097/MPH.0b013e3181d32184. PMID 20186101
- [Background] Wuyts WA, Vanaudenaerde BM, Dupont LJ, Van Raemdonck DE, Demedts MG, Verleden GM. N-acetylcysteine inhibits interleukin-17-induced interleukin-8 production from human airway smooth muscle cells: a possible role for anti-oxidative treatment in chronic lung rejection? J Heart Lung Transplant. 2004 Jan;23(1):122-7. doi: 10.1016/s1053-2498(03)00099-8. PMID 14734137